CLINICAL TRIAL: NCT01684124
Title: A Before-and-after Assessment of Conservative Oxygen Therapy vs. Standard Care in Critically Ill Mechanically Ventilated Patients
Brief Title: An Assessment of the Feasibility and Safety of Conservative Oxygen Therapy in Critically Ill Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Austin Health (Other Government)
Responsible Party: Principal Investigator, Rinaldo Bellomo, Director of ICU Research, Austin Health
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AICU2012-008
Record Dates: First submitted 2012-09-07; First posted 2012-09-12 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Critical Illness
Keywords: oxygen; critical illness; mechanical ventilation
MeSH Terms: conditions — Critical Illness | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- standard care (Placebo Comparator): normal treatment
  Interventions: Other: standard care
- conservative O2 therapy (Active Comparator): a value of 90-92% O2 saturation will be targeted
  Interventions: Other: conservative O2 therapy

INTERVENTIONS:
Other: conservative O2 therapy — target lower O2 saturation
  Arms: conservative O2 therapy
Other: standard care
  Arms: standard care

SUMMARY:
The investigators hypothesize that it is feasible and safe to deliver a conservative approach to oxygen therapy in mechanically ventilated critically ill patients (a tiem frame of, on average,10 days).

DETAILED DESCRIPTION:
1. Identify patients likely to require ventilation until the day after tomorrow (a time frame of 36 hours of average)
2. Deliver a conservative oxygen therapy protocol while in ICU (a time frame on average of 10 days)
3. Target an oxygen saturation between 90 and 92%
4. Adjust FiO2 to achieve target SaO2 at all times
5. Assess percentage of time patient is within target
6. Assess for safety of this approach

ELIGIBILITY:
Inclusion Criteria:

* Mechanical ventilation
* expected to be ventilated until the day after tomorrow (a tiem frame of, on average 48 hours)

Exclusion Criteria:

* expected to be off mechanical ventilation today or tomorrow
* carbon monoxide poisoning
* necrotizing fasciitis

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2012-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Difference in PaO2/FiO2 ratio from baseline to worst value | 10 days
  Pao2/FiO2 ratio will be measured regularly and compared during standard care and the intervention period (a time frame of, on average, 10 days)

SECONDARY OUTCOMES:
Lactate | 10 days
  blood lactate will be measured regularly and assessed during standard care and the intervention period

OTHER OUTCOMES:
arrhythmias | 10 days
  patients will have continuous ECG monitoring and arrhythmias will be recorded in the two groups

CONTACTS AND LOCATIONS:
Locations (1):
- Austin Hospital, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Eastwood GM, Tanaka A, Espinoza ED, Peck L, Young H, Martensson J, Zhang L, Glassford NJ, Hsiao YF, Suzuki S, Bellomo R. Conservative oxygen therapy in mechanically ventilated patients following cardiac arrest: A retrospective nested cohort study. Resuscitation. 2016 Apr;101:108-14. doi: 10.1016/j.resuscitation.2015.11.026. Epub 2015 Dec 21. PMID 26718090